CLINICAL TRIAL: NCT03990766
Title: SCENT Trial: Nasal Theophylline Irrigation for Treatment of Post-Viral Olfactory Dysfunction
Brief Title: Smell Changes & Efficacy of Nasal Theophylline
Acronym: SCENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201901107
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Olfactory Disorder; Anosmia; Viral Infection; Theophylline Causing Adverse Effects in Therapeutic Use; Smell Disorder
Keywords: Olfactory dysfunction; Anosmia; Hyposmia; Post-viral; Theophylline; Adverse effects; Smell
MeSH Terms: conditions — Anosmia; Virus Diseases; Olfaction Disorders | interventions — Theophylline; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Two randomized arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Theophylline saline irrigation (Experimental): Theophylline 12 mg capsule contents dissolved into a sinus rinse bottle containing distilled or boiled tap water and USP Grade Sodium Chloride & Sodium Bicarbonate Mixture commercially prepared packets, delivered to the bilateral nasal cavities twice daily.
  Interventions: Drug: Theophylline
- Placebo saline irrigation (Placebo Comparator): Identical-appearing lactose monohydrate capsule contents dissolved into a sinus rinse bottle containing distilled or boiled tap water and USP Grade Sodium Chloride & Sodium Bicarbonate Mixture commercially prepared packets, delivered to the bilateral nasal cavities twice daily.
  Interventions: Drug: Saline Nasal

INTERVENTIONS:
Drug: Theophylline — Theophylline delivered via high-volume, low-pressure nasal saline irrigation
  Arms: Theophylline saline irrigation
Drug: Saline Nasal — Lactose delivered via high-volume, low-pressure nasal saline irrigation
  Arms: Placebo saline irrigation

SUMMARY:
This study evaluates the efficacy and safety of nasal theophylline irrigation in treating smell loss related to a viral respiratory infection. Half the participants will undergo nasal theophylline irrigation treatment while the other half will undergo placebo nasal irrigation with saline alone. All participants will have their sense of smell tested before and after 6 weeks of treatment. All participants will also be regularly asked about any potential side effects related to treatment. In addition, the first 10 participants will have their blood drawn to measure their theophylline level after 1 week of starting treatment to ensure it is not abnormally elevated.

ELIGIBILITY:
Inclusion Criteria:

* Subjective or clinically diagnosed olfactory dysfunction of 6 months to 36 months duration after a presumed viral upper respiratory infection
* Ability to read, write, and understand English

Exclusion Criteria:

* Dependence on theophylline for comorbid conditions such as asthma and chronic obstructive pulmonary disease
* History of an allergic reaction to theophylline or other methylxanthines
* Prior sinonasal or anterior skull base surgery
* Nasal polyposis
* History of neurodegenerative disease (ie. Alzheimer's dementia, Parkinson's disease, Lewy body dementia, frontotemporal dementia)
* Pregnant or breastfeeding mothers
* Current use of medications with significant (≥40%) interactions with theophylline, which include cimetidine, ciprofloxacin, disulfiram, enoxacin, fluvoxamine, interferon-alpha, lithium, mexiletine, phenytoin, propafenone, propranolol, tacrine, thiabendazole, ticlopidine, and troleandomycin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Theophylline: 12 mg of theophylline dissolved in 240 mL of saline, administered to the bilateral nasal cavities twice a day for 6 weeks
- Placebo: Lactose capsule contents dissolved in 240 mL of saline, administered to the bilateral nasal cavities twice a day for 6 weeks
Period: Overall Study
Arm/Group | Theophylline | Placebo
Started | 14 | 13
Completed | 12 | 10
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theophylline Saline Irrigation | Placebo Saline Irrigation | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Median (Full Range); unit: years] | 57.5 [40 to 70] | 59.5 [32 to 67] | 59.0 [32 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
Body Mass Index [Median (Full Range); unit: kg/m^2] | 32.3 [21.6 to 49.5] | 33.0 [22.7 to 45.6] | 33.0 [21.6 to 49.5]
Smoking history [Count of Participants; unit: Participants] | 0 | 2 | 2
Deviated septum [Count of Participants; unit: Participants] | 3 | 2 | 5
Diabetes mellitus [Count of Participants; unit: Participants] | 1 | 1 | 2
Obstructive sleep apnea on positive airway pressure [Count of Participants; unit: Participants] | 2 | 0 | 2
Hypothyroidism [Count of Participants; unit: Participants] | 3 | 1 | 4
Family history of dementia [Count of Participants; unit: Participants] | 2 | 1 | 3
Moderate/severe comorbidity (ACE-27 scores 2-3) [Count of Participants; unit: Participants] | 5 | 1 | 6
Prior oral steroids [Count of Participants; unit: Participants] | 8 | 6 | 14
Prior nasal steroids [Count of Participants; unit: Participants] | 9 | 7 | 16
Prior olfactory training [Count of Participants; unit: Participants] | 1 | 2 | 3
Time from upper respiratory infection to treatment [Median (Full Range); unit: months] | 11.0 [6.2 to 27.5] | 8.4 [6.4 to 27.6] | 8.8 [6.2 to 27.6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Improvement in Global Rating of Smell Change
Description: Self-reported change in smell after intervention on a 7-point Likert scale. Response options with corresponding point values: 7) Much better, 6) Somewhat better, 5) Slightly better, 4) Neither better nor worse, 3) Slightly worse, 2) Somewhat worse, and 1) Much worse. The maximum score is 7, and higher values indicate better outcomes. A score of 4 is considered neutral. Scores of 5 or higher indicated clinical improvement.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 12 | 10
Participants | 4 | 3
Statistical Analysis 1: Comparison: Theophylline vs Placebo; Test type: Superiority; Risk Difference (RD) = 3.3, 95% CI 2-sided [-35.6 to 42.3]

2. Secondary Outcome: University of Pennsylvania Smell Identification Test (UPSIT) Total Score Change
Description: Within- and between-subject changes in UPSIT total scores measured at baseline and at 6 weeks after therapy. This test is a validated 40-question forced-choice odor identification test where microencapsulated odorants on a strip are released by scratching. Each question corresponds to one point, and there are no subscales. The minimum score is 0 while the maximum score is 40, and higher values indicate better outcomes.
Time Frame: 6 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 12 | 10
score on a scale | 1 [-4 to 12] | 0 [-8 to 5]
Statistical Analysis 1: Comparison: Theophylline vs Placebo; Test type: Superiority; Median Difference (Net) = 1, 95% CI 2-sided [-3 to 5]

3. Secondary Outcome: Questionnaire of Olfactory Disorders-Negative Statements (QOD-NS) Score Change
Description: Within- and between-subject changes in QOD-NS scores measured at baseline and at 6 weeks after therapy, which is a validated 17-item questionnaire about quality of life and impairments related to olfactory dysfunction. Each question is scored from 0 to 3 points, and there are no subscales. The minimum score is 0 while the maximum score is 51, and higher values indicate worse quality of life or higher degree of impairment.
Time Frame: 6 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 12 | 10
score on a scale | -6.5 [-15 to 4] | 1.5 [-4 to 19]
Statistical Analysis 1: Comparison: Theophylline vs Placebo; The within-subject change in QOD-NS scores from baseline and 6 weeks was calculated for each individual patient. Then the median of all the patients' change in score for each cohort was calculated. Because these were within-subject changes in scores, the median difference values for each cohort do not necessarily correspond with simply subtracting the median change in score in the theophylline cohort from the median change in score in the placebo cohort; Test type: Superiority; Median Difference (Net) = -10, 95% CI 2-sided [-15 to -4]

4. Secondary Outcome: Olfactory Dysfunction Outcomes Ratings (ODOR) Score Change
Description: Within- and between-subject changes measured at baseline and at 6 weeks after therapy. This test is a new disease-specific 28-item questionnaire that assesses for physical, functional, and emotional limitations in patients with olfactory dysfunction of any etiology. Each question is scored from 0 to 4. The minimum score is 0 while the maximum score is 112, and higher values indicate higher degree of limitations and worse outcomes. There are no subscales within the current questionnaire.
Time Frame: 6 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 12 | 10
score on a scale | -1.5 [-18 to 6] | -7.5 [-29 to 6]
Statistical Analysis 1: Comparison: Theophylline vs Placebo; The within-subject change in ODOR scores from baseline and 6 weeks was calculated for each individual patient. Then the median of all the patients' change in score for each cohort was calculated. Because these were within-subject changes in scores, the median difference values for each cohort do not necessarily correspond with simply subtracting the median change in score in the theophylline cohort from the median change in score in the placebo cohort. We confirmed the reported results; Test type: Superiority; Median Difference (Net) = 7, 95% CI 2-sided [-2 to 17]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 6 weeks of treatment
Description: The first 10 participants regardless of intervention underwent theophylline level measurements after 1 week of treatment. If a measurable amount of theophylline was identified, the test would be immediately repeated. If theophylline was detected in the second sample, the plan was to continue measuring in another 10 subjects. In addition, all participants were queried biweekly regarding any adverse effects.
Arm/Group | Theophylline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Theophylline (N=14) | Placebo (N=13)
Detectable serum theophylline (Blood and lymphatic system disorders) | 0/5 (0) | 0/5 (0) — Detectable serum theophylline level measured by phlebotomy after 1 week of treatment in the first 10 patients

LIMITATIONS AND CAVEATS:
The diagnosis of PVOD is by patient history and is thus subject to recall bias. In addition, PVOD treatment response may differ according to the causative virus, which is rarely known. The sample size was limited since all non-life saving clinical research and recruitment were halted at our institution at the time due to COVID-19. Lastly, the optimal dosing of theophylline irrigations is yet to be determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT03990766/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT03990766/ICF_001.pdf